CLINICAL TRIAL: NCT00160615
Title: Follow-up Study of L059 (Levetiracetam) in Epileptic Patients With Partial Onset Seizures by Open Label Method
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01020
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy, partial; Keppra; Levetiracetam
MeSH Terms: conditions — Epilepsies, Partial | interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: This study N01020 (NCT00160615) was designed as a single group assignment study and as follow-up study, open for patients from N165 (NCT00600509). The differentiation into placebo and Levetiracetam in the results reporting section is based on the treatment of the previously conducted study N165 (NCT00600509).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Levetiracetam (Experimental): Subjects received oral tablets of Levetiracetam. This study N01020 (NCT00160615) was designed as a single group assignment study and as follow-up study, open for patients from N165 (NCT00600509). The differentiation into placebo and Levetiracetam in the results reporting section is based on the treatment of the previously conducted study N165 (NCT00600509).
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — * Pharmaceutical form: Film-coating tablets
  * Concentration: 250 mg/ 500 mg
  * Route of administration: oral use
  Other Names: Keppra

SUMMARY:
The safety and efficacy of L059 was evaluated in patients who completed "N165 Clinical Trial of L059". They received L059 at a daily dose from 1,000 mg to 3,000 mg in addition to their standard concomitant AEDs

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the evaluation period (Week 16) of N165 Clinical Trial of L059
* Patients/the parent or guardian wish to continue treatment with L059 and to enter N165 Follow-up Study, and also the investigator admit the necessity of the repeated intake of the investigational drug for the patients.

Exclusion Criteria:

* Patients who had not participate in N165 Clinical Trial of L059.
* Patients who had participated in N165 Clinical Trial of L059 with no intention of entering the follow-up study taking the same medication.
* Patients had not been in compliance with requirements of Protocol for N165 Clinical Trial of L059 in the course of the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2001-09-12 (Actual); Primary Completion 2007-01-17 (Actual); Study Completion 2007-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in September 2001 and concluded in January 2007.
Pre-assignment Details: Participant Flow refers to the Full Analysis Set (FAS). Of the 154 subjects who enrolled in the study, 151 subjects were included in the FAS population and 3 subjects were identified with major protocol deviations leading to exclusion from FAS.
Groups:
- N165 Randomized Treatment PBO: Subjects received Placebo (PBO) in study N165 [NCT00600509] and received LEV in this study: After starting with the 4 week-fixed 3000 mg/day, the daily doses of LEV were permitted to be adjusted by 500 or 1000 mg/day at a 4-week interval between 1000 mg/day and 3000 mg/day.
- N165 Randomized Treatment LEV: Subjects received Levetiracetam (LEV) in study N165 [NCT00600509] and received LEV in this study: After starting with the 4 week-fixed 3000 mg/day, the daily doses of LEV were permitted to be adjusted by 500 or 1000 mg/day at a 4-week interval between 1000 mg/day and 3000 mg/day.
Period: Overall Study
Arm/Group | N165 Randomized Treatment PBO | N165 Randomized Treatment LEV
Started | 50 | 101
Completed | 32 | 56
Not Completed | 18 | 45
Not completed — Adverse Event | 5 | 12
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 11 | 23
Not completed — Patient decision | 1 | 2
Not completed — Investigator decision | 1 | 1
Not completed — AE agents had to be discontinued (exam.) | 0 | 1
Not completed — Switch to surgical treatment | 0 | 2
Not completed — Non-compliance was suspected | 0 | 1
Not completed — Poor compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis Set (FAS)
Groups:
- N165 Randomized Treatment PBO (FAS): Subjects received Placebo (PBO) in study N165 [NCT00600509] and received LEV in this study: After starting with the 4 week-fixed 3000 mg/day, the daily doses of LEV were permitted to be adjusted by 500 or 1000 mg/day at a 4-week interval between 1000 mg/day and 3000 mg/day.
- N165 Randomized Treatment LEV (FAS): Subjects received Levetiracetam (LEV) in study N165 [NCT00600509] and received LEV in this study: After starting with the 4 week-fixed 3000 mg/day, the daily doses of LEV were permitted to be adjusted by 500 or 1000 mg/day at a 4-week interval between 1000 mg/day and 3000 mg/day.
Arm/Group | N165 Randomized Treatment PBO (FAS) | N165 Randomized Treatment LEV (FAS) | Total Title
Number analyzed (Participants) | 50 | 101 | 151
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.19 (9.99) | 31.95 (10.19) | 32.36 (10.11)
Age, Customized [Number; unit: Participants]
  <=18 years | 2 | 6 | 8
  Between 18 and 65 years | 48 | 95 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 47 | 74
  Male | 23 | 54 | 77

OUTCOME MEASURES:

1. Primary Outcome: Partial (Type I) Seizure Frequency Per Week by Analysis Visit
Description: Number of Partial (Type I) seizures over the treatment period standardized to 1 week period.
Time Frame: From Baseline up to 54 months
Population: Full Analysis set included 151 subjects. Only subjects with valid data for partial (Type I) seizure frequency per week at the respective visit are included in the analysis. Number of participants analyzed is given separately per visit.
Measure: Median (Inter-Quartile Range); unit: Number of Seizures (Type I) per week
Arm/Group | N165 Randomized Treatment PBO | N165 Randomized Treatment LEV
Number analyzed (Participants) | 50 | 101
Number of Seizures (Type I) per week
  >= 1 day(d) - <= 3 months(m): number analyzed (Participants) | 50 | 100
  >= 1 day(d) - <= 3 months(m) | 1.68 [1.18 to 4.06] | 2.19 [0.99 to 5.41]
  > 3 m - <= 6 m: number analyzed (Participants) | 43 | 92
  > 3 m - <= 6 m | 1.69 [1.00 to 2.75] | 2.00 [0.87 to 4.48]
  > 6 m - <= 9 m: number analyzed (Participants) | 40 | 82
  > 6 m - <= 9 m | 1.58 [0.88 to 2.69] | 1.78 [0.68 to 4.94]
  > 9 m - <= 12 m: number analyzed (Participants) | 39 | 78
  > 9 m - <= 12 m | 1.41 [0.95 to 3.25] | 1.60 [0.60 to 5.05]
  > 12 m - <= 15 m: number analyzed (Participants) | 35 | 68
  > 12 m - <= 15 m | 1.58 [1.06 to 2.50] | 1.55 [0.80 to 4.67]
  > 15 m - <= 18 m: number analyzed (Participants) | 32 | 64
  > 15 m - <= 18 m | 1.36 [1.03 to 2.32] | 1.69 [0.75 to 4.80]
  > 18 m - <= 21 m: number analyzed (Participants) | 30 | 61
  > 18 m - <= 21 m | 1.35 [0.72 to 1.96] | 1.51 [0.62 to 4.49]
  > 21 m - <= 24 m: number analyzed (Participants) | 30 | 59
  > 21 m - <= 24 m | 1.30 [0.75 to 1.98] | 1.36 [0.67 to 3.17]
  > 24 m - <= 27 m: number analyzed (Participants) | 30 | 56
  > 24 m - <= 27 m | 1.25 [0.56 to 2.38] | 1.33 [0.82 to 2.80]
  > 27 m - <= 30 m: number analyzed (Participants) | 30 | 55
  > 27 m - <= 30 m | 1.30 [0.66 to 2.46] | 1.28 [0.72 to 2.75]
  > 30 m - <= 33 m: number analyzed (Participants) | 29 | 52
  > 30 m - <= 33 m | 1.21 [0.71 to 2.65] | 1.33 [0.77 to 2.83]
  > 33 m - <= 36 m: number analyzed (Participants) | 29 | 49
  > 33 m - <= 36 m | 1.14 [0.68 to 2.69] | 1.30 [0.71 to 3.31]
  > 36 m - <= 39 m: number analyzed (Participants) | 28 | 49
  > 36 m - <= 39 m | 1.20 [0.65 to 2.92] | 1.28 [0.75 to 3.32]
  > 39 m - <= 42 m: number analyzed (Participants) | 27 | 43
  > 39 m - <= 42 m | 1.25 [0.50 to 2.91] | 1.32 [0.58 to 2.62]
  > 42 m - <= 45 m: number analyzed (Participants) | 20 | 30
  > 42 m - <= 45 m | 1.17 [0.79 to 2.41] | 1.28 [0.60 to 2.49]
  > 45 m - <= 48 m: number analyzed (Participants) | 16 | 23
  > 45 m - <= 48 m | 0.95 [0.54 to 2.05] | 1.09 [0.25 to 1.58]
  > 48 m - <= 51 m: number analyzed (Participants) | 12 | 17
  > 48 m - <= 51 m | 0.90 [0.31 to 1.61] | 0.70 [0.14 to 1.42]
  > 51 m - <= 54 m: number analyzed (Participants) | 10 | 12
  > 51 m - <= 54 m | 1.06 [0.08 to 2.17] | 0.78 [0.11 to 1.33]
  > 54 m: number analyzed (Participants) | 8 | 5
  > 54 m | 1.16 [0.27 to 1.65] | 0.09 [0.08 to 1.16]

2. Primary Outcome: Partial (Type IA) Seizure Frequency Per Week by Analysis Visit
Description: Number of Partial (Type IA) seizures over the treatment period standardized to 1 week period.
Time Frame: From Baseline up to 54 months
Population: Subjects with Type IA seizure count equal to zero during baseline and evaluation periods are excluded. Only subjects with valid data for partial (Type IA) seizure frequency per week at the respective visit are included in the analysis. Number of participants analyzed is given separately per visit.
Measure: Median (Inter-Quartile Range); unit: Number of Seizures (Type IA) per week
Arm/Group | N165 Randomized Treatment PBO | N165 Randomized Treatment LEV
Number analyzed (Participants) | 23 | 61
Number of Seizures (Type IA) per week
  >= 1 d - <= 3 m: number analyzed (Participants) | 23 | 60
  >= 1 d - <= 3 m | 0.86 [0.07 to 1.73] | 0.68 [0.06 to 4.41]
  > 3 m - <= 6 m: number analyzed (Participants) | 20 | 58
  > 3 m - <= 6 m | 0.32 [0.06 to 1.44] | 0.83 [0.06 to 3.31]
  > 6 m - <= 9 m: number analyzed (Participants) | 18 | 53
  > 6 m - <= 9 m | 0.24 [0.00 to 1.33] | 0.63 [0.05 to 4.67]
  > 9 m - <= 12 m: number analyzed (Participants) | 18 | 51
  > 9 m - <= 12 m | 0.26 [0.00 to 1.23] | 0.50 [0.00 to 3.47]
  > 12 m - <= 15 m: number analyzed (Participants) | 16 | 44
  > 12 m - <= 15 m | 0.57 [0.09 to 1.35] | 0.22 [0.00 to 2.74]
  > 15 m - <= 18 m: number analyzed (Participants) | 15 | 43
  > 15 m - <= 18 m | 0.27 [0.00 to 1.32] | 0.30 [0.00 to 2.81]
  > 18 m - <= 21 m: number analyzed (Participants) | 13 | 41
  > 18 m - <= 21 m | 0.10 [0.00 to 1.38] | 0.42 [0.00 to 1.82]
  > 21 m - <= 24 m: number analyzed (Participants) | 13 | 39
  > 21 m - <= 24 m | 0.17 [0.06 to 1.00] | 0.43 [0.05 to 1.60]
  > 24 m - <= 27 m: number analyzed (Participants) | 13 | 36
  > 24 m - <= 27 m | 0.29 [0.00 to 1.10] | 0.25 [0.00 to 1.41]
  > 27 m - <= 30 m: number analyzed (Participants) | 13 | 34
  > 27 m - <= 30 m | 0.44 [0.00 to 1.06] | 0.17 [0.00 to 1.41]
  > 30 m - <= 33 m: number analyzed (Participants) | 13 | 33
  > 30 m - <= 33 m | 0.24 [0.00 to 0.98] | 0.25 [0.08 to 1.32]
  > 33 m - <= 36 m: number analyzed (Participants) | 13 | 31
  > 33 m - <= 36 m | 0.17 [0.00 to 0.83] | 0.29 [0.05 to 1.63]
  > 36 m - <= 39 m: number analyzed (Participants) | 13 | 31
  > 36 m - <= 39 m | 0.14 [0.00 to 0.40] | 0.13 [0.04 to 1.50]
  > 39 m - <= 42 m: number analyzed (Participants) | 12 | 28
  > 39 m - <= 42 m | 0.17 [0.00 to 0.83] | 0.28 [0.04 to 1.29]
  > 42 m - <= 45 m: number analyzed (Participants) | 11 | 20
  > 42 m - <= 45 m | 0.09 [0.00 to 1.13] | 0.44 [0.08 to 1.03]
  > 45 m - <= 48 m: number analyzed (Participants) | 8 | 16
  > 45 m - <= 48 m | 0.20 [0.08 to 0.97] | 0.48 [0.09 to 1.38]
  > 48 m - <= 51 m: number analyzed (Participants) | 6 | 11
  > 48 m - <= 51 m | 0.44 [0.00 to 1.42] | 0.18 [0.00 to 1.17]
  > 51 m - <= 54 m: number analyzed (Participants) | 5 | 9
  > 51 m - <= 54 m | 0.62 [0.00 to 1.59] | 0.17 [0.10 to 0.63]
  > 54 m: number analyzed (Participants) | 4 | 5
  > 54 m | 0.87 [0.14 to 1.65] | 0.08 [0.00 to 0.84]

3. Primary Outcome: Partial (Type IB) Seizure Frequency Per Week by Analysis Visit
Description: Number of Partial (Type IB) seizures over the treatment period standardized to 1 week period.
Time Frame: From Baseline up to 54 months
Population: Subjects with Type IB seizure count equal to zero during baseline and evaluation periods are excluded. Only subjects with valid data for partial (Type IB) seizure frequency per week at the respective visit are included in the analysis. Number of participants analyzed is given separately per visit.
Measure: Median (Inter-Quartile Range); unit: Number of Seizures (Type IB) per week
Arm/Group | N165 Randomized Treatment PBO | N165 Randomized Treatment LEV
Number analyzed (Participants) | 44 | 91
Number of Seizures (Type IB) per week
  >= 1 d - <= 3 m: number analyzed (Participants) | 43 | 91
  >= 1 d - <= 3 m | 1.56 [0.94 to 2.49] | 1.27 [0.50 to 3.25]
  > 3 m - <= 6 m: number analyzed (Participants) | 37 | 83
  > 3 m - <= 6 m | 1.51 [0.81 to 2.69] | 1.13 [0.38 to 3.18]
  > 6 m <= 9 m: number analyzed (Participants) | 34 | 74
  > 6 m <= 9 m | 1.30 [0.60 to 2.25] | 0.92 [0.25 to 2.31]
  > 9 m - <= 12 m: number analyzed (Participants) | 33 | 71
  > 9 m - <= 12 m | 1.39 [0.80 to 1.88] | 0.72 [0.24 to 2.11]
  > 12 m - <= 15 m: number analyzed (Participants) | 30 | 62
  > 12 m - <= 15 m | 1.34 [0.71 to 1.94] | 0.81 [0.38 to 2.12]
  > 15 m - <= 18 m: number analyzed (Participants) | 27 | 58
  > 15 m - <= 18 m | 1.25 [0.81 to 2.21] | 0.81 [0.35 to 1.88]
  > 18 m - <= 21 m: number analyzed (Participants) | 25 | 56
  > 18 m - <= 21 m | 1.25 [0.72 to 1.95] | 0.58 [0.31 to 2.34]
  > 21 m - <= 24 m: number analyzed (Participants) | 25 | 54
  > 21 m - <= 24 m | 1.26 [0.70 to 1.90] | 0.73 [0.26 to 2.65]
  > 24 m - <= 27 m: number analyzed (Participants) | 25 | 52
  > 24 m - <= 27 m | 1.21 [0.56 to 2.50] | 0.85 [0.13 to 2.05]
  > 27 m - <= 30 m: number analyzed (Participants) | 25 | 52
  > 27 m - <= 30 m | 1.21 [0.66 to 3.33] | 0.98 [0.15 to 1.74]
  > 30 m - <= 33 m: number analyzed (Participants) | 24 | 50
  > 30 m - <= 33 m | 1.25 [0.69 to 2.84] | 0.79 [0.20 to 2.04]
  > 33 m - <= 36 m: number analyzed (Participants) | 24 | 47
  > 33 m - <= 36 m | 1.15 [0.76 to 2.91] | 0.96 [0.14 to 2.13]
  > 36 m - <= 39 m: number analyzed (Participants) | 23 | 47
  > 36 m - <= 39 m | 1.28 [0.80 to 3.43] | 1.04 [0.17 to 2.48]
  > 39 m - <= 42 m: number analyzed (Participants) | 22 | 42
  > 39 m - <= 42 m | 1.40 [0.66 to 3.48] | 0.77 [0.13 to 1.71]
  > 42 m - <= 45 m: number analyzed (Participants) | 16 | 29
  > 42 m - <= 45 m | 1.22 [0.76 to 2.79] | 0.89 [0.08 to 1.52]
  > 45 m - <= 48 m: number analyzed (Participants) | 12 | 22
  > 45 m - <= 48 m | 0.87 [0.46 to 2.89] | 0.27 [0.00 to 1.36]
  > 48 m - <= 51 m: number analyzed (Participants) | 8 | 16
  > 48 m - <= 51 m | 0.74 [0.33 to 2.46] | 0.22 [0.02 to 1.15]
  > 51 m - <= 54 m: number analyzed (Participants) | 6 | 12
  > 51 m - <= 54 m | 0.80 [0.46 to 3.64] | 0.19 [0.00 to 1.25]
  > 54 m: number analyzed (Participants) | 5 | 5
  > 54 m | 0.72 [0.54 to 1.33] | 0.09 [0.00 to 0.17]

4. Primary Outcome: Partial (Type IC) Seizure Frequency Per Week by Analysis Visit
Description: Number of Partial (Type IC) seizures over the treatment period standardized to 1 week period.
Time Frame: From Baseline up to 54 months
Population: Subjects with Type IC seizure count equal to zero during baseline and evaluation periods are excluded. Only subjects with valid data for partial (Type IC) seizure frequency per week at the respective visit are included in the analysis. Number of participants analyzed is given separately per visit.
Measure: Median (Inter-Quartile Range); unit: Number of Seizures (Type IC) per week
Arm/Group | N165 Randomized Treatment PBO | N165 Randomized Treatment LEV
Number analyzed (Participants) | 18 | 42
Number of Seizures (Type IC) per week
  >= 1 d - <= 3 m: number analyzed (Participants) | 18 | 40
  >= 1 d - <= 3 m | 0.00 [0.00 to 0.31] | 0.00 [0.00 to 0.19]
  > 3 m - <= 6 m: number analyzed (Participants) | 15 | 39
  > 3 m - <= 6 m | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 0.07]
  > 6 m - <= 9 m: number analyzed (Participants) | 14 | 37
  > 6 m - <= 9 m | 0.05 [0.00 to 0.19] | 0.00 [0.00 to 0.13]
  > 9 m - <= 12 m: number analyzed (Participants) | 14 | 37
  > 9 m - <= 12 m | 0.06 [0.00 to 0.17] | 0.00 [0.00 to 0.06]
  > 12 m - <= 15 m: number analyzed (Participants) | 14 | 32
  > 12 m - <= 15 m | 0.06 [0.00 to 0.07] | 0.00 [0.00 to 0.03]
  > 15 m - <= 18 m: number analyzed (Participants) | 13 | 30
  > 15 m - <= 18 m | 0.00 [0.00 to 0.13] | 0.00 [0.00 to 0.06]
  > 18 m - <= 21 m: number analyzed (Participants) | 11 | 29
  > 18 m - <= 21 m | 0.00 [0.00 to 0.17] | 0.00 [0.00 to 0.00]
  > 21 m - <= 24 m: number analyzed (Participants) | 10 | 26
  > 21 m - <= 24 m | 0.05 [0.00 to 0.14] | 0.00 [0.00 to 0.00]
  > 24 m - <= 27 m: number analyzed (Participants) | 10 | 25
  > 24 m - <= 27 m | 0.02 [0.00 to 0.17] | 0.00 [0.00 to 0.00]
  > 27 m - <= 30 m: number analyzed (Participants) | 11 | 26
  > 27 m - <= 30 m | 0.04 [0.00 to 0.13] | 0.00 [0.00 to 0.00]
  > 30 m - <= 33 m: number analyzed (Participants) | 10 | 25
  > 30 m - <= 33 m | 0.09 [0.00 to 0.16] | 0.00 [0.00 to 0.00]
  > 33 m - <= 36 m: number analyzed (Participants) | 10 | 25
  > 33 m - <= 36 m | 0.06 [0.00 to 0.13] | 0.00 [0.00 to 0.00]
  > 36 m - <= 39 m: number analyzed (Participants) | 10 | 25
  > 36 m - <= 39 m | 0.04 [0.00 to 0.08] | 0.00 [0.00 to 0.00]
  > 39 m - <= 42 m: number analyzed (Participants) | 9 | 22
  > 39 m - <= 42 m | 0.08 [0.00 to 0.08] | 0.00 [0.00 to 0.00]
  > 42 m - <= 45 m: number analyzed (Participants) | 8 | 12
  > 42 m - <= 45 m | 0.04 [0.00 to 0.19] | 0.00 [0.00 to 0.02]
  > 45 m - <= 48 m: number analyzed (Participants) | 6 | 9
  > 45 m - <= 48 m | 0.02 [0.00 to 0.04] | 0.00 [0.00 to 0.00]
  > 48 m - <= 51 m: number analyzed (Participants) | 5 | 7
  > 48 m - <= 51 m | 0.00 [0.00 to 0.04] | 0.00 [0.00 to 0.00]
  > 51 m - <= 54 m: number analyzed (Participants) | 5 | 4
  > 51 m - <= 54 m | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  > 54 m: number analyzed (Participants) | 3 | 1
  > 54 m | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

5. Secondary Outcome: Percentage Change From Baseline of Partial Onset Seizure Frequency (Type I Overall) Per Week by Analysis Visit
Description: Percentage change from baseline of of Partial (Type I) seizure frequency over the treatment period standardized to 1 week period.
  Negative values indicate improvement from Baseline.
Time Frame: From Baseline up to 54 months
Population: Full Analysis set included 151 subjects. Only subjects with valid data for Partial (Type I seizure frequency per week at the respective visit are included in the analysis. Number of participants analyzed is given separately per visit.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | N165 Randomized Treatment PBO | N165 Randomized Treatment LEV
Number analyzed (Participants) | 50 | 101
Percent change
  >= 1 d - <= 3 m: number analyzed (Participants) | 50 | 100
  >= 1 d - <= 3 m | -27.39 [-48.11 to 5.37] | -31.24 [-61.33 to 2.86]
  > 3 m - <= 6 m: number analyzed (Participants) | 43 | 92
  > 3 m - <= 6 m | -35.15 [-58.61 to -6.20] | -34.74 [-62.48 to -3.22]
  > 6 m - <= 9 m: number analyzed (Participants) | 40 | 82
  > 6 m - <= 9 m | -38.42 [-59.44 to 5.08] | -43.03 [-77.38 to -9.61]
  > 9 m - <= 12 m: number analyzed (Participants) | 39 | 78
  > 9 m - <= 12 m | -41.44 [-61.30 to -6.63] | -43.11 [-73.76 to -11.60]
  > 12 m - <= 15 m: number analyzed (Participants) | 35 | 68
  > 12 m - <= 15 m | -29.58 [-58.69 to -10.04] | -46.38 [-73.80 to -11.12]
  > 15 m - <= 18 m: number analyzed (Participants) | 32 | 64
  > 15 m - <= 18 m | -44.44 [-70.68 to -19.37] | -43.17 [-69.33 to -16.84]
  > 18 m - <= 21 m: number analyzed (Participants) | 30 | 61
  > 18 m - <= 21 m | -37.58 [-69.96 to -21.23] | -49.61 [-71.95 to -20.04]
  > 21 m - <= 24 m: number analyzed (Participants) | 30 | 59
  > 21 m - <= 24 m | -45.75 [-59.76 to -15.74] | -52.96 [-77.16 to -13.78]
  > 24 m - <= 27 m: number analyzed (Participants) | 30 | 56
  > 24 m - <= 27 m | -50.89 [-69.36 to 0.01] | -53.78 [-73.22 to -23.05]
  > 27 m - <= 30 m: number analyzed (Participants) | 30 | 55
  > 27 m - <= 30 m | -40.54 [-74.09 to -1.74] | -47.71 [-76.29 to -18.07]
  > 30 m - <= 33 m: number analyzed (Participants) | 29 | 52
  > 30 m - <= 33 m | -29.96 [-69.05 to 0.00] | -43.09 [-76.80 to -16.09]
  > 33 m - <= 36 m: number analyzed (Participants) | 29 | 49
  > 33 m - <= 36 m | -40.03 [-72.14 to -5.33] | -39.01 [-75.01 to -11.31]
  > 36 m - <= 39 m: number analyzed (Participants) | 28 | 49
  > 36 m - <= 39 m | -43.67 [-68.70 to 3.89] | -44.42 [-74.06 to -9.63]
  > 39 m - <= 42 m: number analyzed (Participants) | 27 | 43
  > 39 m - <= 42 m | -42.88 [-65.68 to 0.20] | -47.69 [-85.88 to -10.34]
  > 42 m - <= 45 m: number analyzed (Participants) | 20 | 30
  > 42 m - <= 45 m | -45.06 [-57.76 to -21.01] | -71.96 [-85.97 to -21.29]
  > 45 m - <= 48 m: number analyzed (Participants) | 16 | 23
  > 45 m - <= 48 m | -42.41 [-71.81 to -28.73] | -80.02 [-86.42 to -36.37]
  > 48 m - <= 51 m: number analyzed (Participants) | 12 | 17
  > 48 m - <= 51 m | -49.11 [-74.26 to -23.92] | -78.28 [-88.06 to -55.91]
  > 51 m - <= 54 m: number analyzed (Participants) | 10 | 12
  > 51 m - <= 54 m | -43.74 [-96.55 to 0.60] | -81.81 [-92.97 to -66.12]
  > 54 m: number analyzed (Participants) | 8 | 5
  > 54 m | -40.72 [-76.94 to -14.12] | -90.00 [-92.17 to -85.37]

6. Secondary Outcome: Percentage Change From Baseline of Partial Onset Seizure Frequency (Subtype IA) Per Week by Analysis Visit
Description: Percentage change from baseline of of Partial (Type IA) seizure frequency over the treatment period standardized to 1 week period.
  Negative values indicate improvement from Baseline.
Time Frame: From Baseline up to 54 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | N165 Randomized Treatment PBO (FAS) | N165 Randomized Treatment LEV (FAS)
Number analyzed (Participants) | 23 | 61
Percent change
  >= 1 d - <= 3 m: number analyzed (Participants) | 22 | 51
  >= 1 d - <= 3 m | -79.58 [-89.22 to -24.55] | -45.93 [-88.28 to 14.97]
  > 3 m - <= 6 m: number analyzed (Participants) | 19 | 49
  > 3 m - <= 6 m | -77.15 [-95.81 to -43.42] | -58.81 [-83.66 to 9.91]
  > 6 m - <= 9 m: number analyzed (Participants) | 17 | 44
  > 6 m - <= 9 m | -71.71 [-100.00 to -39.06] | -61.62 [-86.96 to 45.98]
  > 9 m - <= 12 m: number analyzed (Participants) | 17 | 42
  > 9 m - <= 12 m | -66.05 [-100.00 to -42.98] | -69.01 [-99.09 to -24.55]
  > 12 m - <= 15 m: number analyzed (Participants) | 15 | 37
  > 12 m - <= 15 m | -37.32 [-96.72 to -19.64] | -78.44 [-100.00 to -43.42]
  > 15 m - <= 18 m: number analyzed (Participants) | 14 | 35
  > 15 m - <= 18 m | -79.55 [-100.00 to -46.11] | -71.42 [-93.19 to -9.46]
  > 18 m - <= 21 m: number analyzed (Participants) | 12 | 34
  > 18 m - <= 21 m | -83.68 [-100.00 to -39.59] | -66.07 [-97.31 to -19.52]
  > 21 m - <= 24 m: number analyzed (Participants) | 12 | 34
  > 21 m - <= 24 m | -82.30 [-99.71 to -50.87] | -73.18 [-87.28 to -7.74]
  > 24 m - <= 27 m: number analyzed (Participants) | 12 | 31
  > 24 m - <= 27 m | -72.52 [-99.68 to -49.91] | -74.85 [-91.27 to -33.43]
  > 27 m - <= 30 m: number analyzed (Participants) | 12 | 29
  > 27 m - <= 30 m | -74.89 [-98.71 to -46.15] | -76.45 [-95.81 to -12.09]
  > 30 m - <= 33 m: number analyzed (Participants) | 12 | 29
  > 30 m - <= 33 m | -80.89 [-98.97 to -48.35] | -78.24 [-89.74 to -4.31]
  > 33 m - <= 36 m: number analyzed (Participants) | 12 | 27
  > 33 m - <= 36 m | -84.13 [-100.00 to -48.15] | -80.40 [-96.99 to 9.85]
  > 36 m - <= 39 m: number analyzed (Participants) | 12 | 27
  > 36 m - <= 39 m | -90.62 [-100.00 to -53.87] | -76.79 [-97.71 to -27.78]
  > 39 m - <= 42 m: number analyzed (Participants) | 11 | 24
  > 39 m - <= 42 m | -92.50 [-100.00 to -42.88] | -75.66 [-96.10 to -18.07]
  > 42 m - <= 45 m: number analyzed (Participants) | 10 | 19
  > 42 m - <= 45 m | -77.00 [-99.57 to -47.52] | -74.09 [-93.06 to -39.64]
  > 45 m - <= 48 m: number analyzed (Participants) | 7 | 16
  > 45 m - <= 48 m | -71.43 [-91.25 to -47.31] | -79.25 [-95.95 to -41.45]
  > 48 m - <= 51 m: number analyzed (Participants) | 5 | 11
  > 48 m - <= 51 m | -54.01 [-95.64 to -48.88] | -91.41 [-100.00 to -56.26]
  > 51 m - <= 54 m: number analyzed (Participants) | 5 | 9
  > 51 m - <= 54 m | -64.18 [-100.00 to -42.73] | -83.37 [-98.18 to -71.43]
  > 54 m: number analyzed (Participants) | 4 | 5
  > 54 m | -59.19 [-92.21 to -32.87] | -97.55 [-100.00 to -85.71]

7. Secondary Outcome: Percentage Change From Baseline of Partial Onset Seizure Frequency (Subtype IB) Per Week by Analysis Visit
Description: Percentage change from baseline of of Partial (Type IB) seizure frequency over the treatment period standardized to 1 week period.
  Negative values indicate improvement from Baseline.
Time Frame: From Baseline up to 54 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | N165 Randomized Treatment PBO (FAS) | N165 Randomized Treatment LEV (FAS)
Number analyzed (Participants) | 44 | 91
Percent change
  >= 1 d - <= 3 m: number analyzed (Participants) | 43 | 87
  >= 1 d - <= 3 m | -21.41 [-48.68 to 19.61] | -26.77 [-57.30 to 6.25]
  > 3 m - <= 6 m: number analyzed (Participants) | 37 | 79
  > 3 m - <= 6 m | -21.95 [-52.22 to 2.27] | -31.35 [-64.47 to 0.53]
  > 6 m - <= 9 m: number analyzed (Participants) | 34 | 71
  > 6 m - <= 9 m | -28.30 [-52.22 to 7.30] | -47.61 [-75.99 to -7.14]
  > 9 m - <= 12 m: number analyzed (Participants) | 33 | 67
  > 9 m - <= 12 m | -34.97 [-50.02 to 17.70] | -43.56 [-73.35 to -14.31]
  > 12 m - <= 15 m: number analyzed (Participants) | 30 | 59
  > 12 m - <= 15 m | -21.12 [-54.73 to 7.78] | -51.20 [-74.85 to 6.18]
  > 15 m - <= 18 m: number analyzed (Participants) | 27 | 55
  > 15 m - <= 18 m | -33.18 [-56.67 to 6.88] | -45.80 [-66.80 to -12.59]
  > 18 m - <= 21 m: number analyzed (Participants) | 25 | 53
  > 18 m - <= 21 m | -32.78 [-54.73 to 2.63] | -52.04 [-72.79 to -15.92]
  > 21 m - <= 24 m: number analyzed (Participants) | 25 | 51
  > 21 m - <= 24 m | -20.12 [-58.09 to 1.17] | -52.96 [-78.82 to -10.93]
  > 24 m - <= 27 m: number analyzed (Participants) | 25 | 49
  > 24 m - <= 27 m | -28.75 [-61.84 to 13.15] | -49.71 [-72.31 to -17.12]
  > 27 m - <= 30 m: number analyzed (Participants) | 25 | 49
  > 27 m - <= 30 m | -8.84 [-51.80 to 3.05] | -48.18 [-79.29 to -21.93]
  > 30 m - <= 33 m: number analyzed (Participants) | 24 | 47
  > 30 m - <= 33 m | -15.85 [-52.14 to 16.16] | -46.86 [-79.88 to -11.48]
  > 33 m - <= 36 m: number analyzed (Participants) | 24 | 44
  > 33 m - <= 36 m | -11.73 [-53.45 to 17.68] | -42.03 [-74.93 to -6.07]
  > 36 m - <= 39 m: number analyzed (Participants) | 23 | 44
  > 36 m - <= 39 m | -15.06 [-49.40 to 28.76] | -46.25 [-76.15 to 7.85]
  > 39 m - <= 42 m: number analyzed (Participants) | 22 | 39
  > 39 m - <= 42 m | -20.13 [-53.31 to 31.25] | -49.85 [-86.73 to 0.00]
  > 42 m - <= 45 m: number analyzed (Participants) | 16 | 27
  > 42 m - <= 45 m | -23.76 [-46.47 to 13.76] | -46.51 [-91.95 to -11.07]
  > 45 m - <= 48 m: number analyzed (Participants) | 12 | 20
  > 45 m - <= 48 m | -37.52 [-56.10 to -13.36] | -54.05 [-98.11 to -16.56]
  > 48 m - <= 51 m: number analyzed (Participants) | 8 | 15
  > 48 m - <= 51 m | -42.17 [-53.57 to 1.70] | -77.08 [-94.99 to -38.37]
  > 51 m - <= 54 m: number analyzed (Participants) | 6 | 11
  > 51 m - <= 54 m | 5.38 [-44.75 to 10.33] | -74.58 [-100.00 to 42.13]
  > 54 m: number analyzed (Participants) | 5 | 4
  > 54 m | 3.55 [-47.49 to 74.45] | -86.61 [-93.85 to -8.06]

8. Secondary Outcome: Percentage Change From Baseline of Partial Onset Seizure Frequency (Subtype IC) Per Week by Analysis Visit
Description: Percentage change from baseline of of Partial (Type IC) seizure frequency over the treatment period standardized to 1 week period.
  Negative values indicate improvement from Baseline.
Time Frame: From Baseline up to 54 months
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | N165 Randomized Treatment PBO | N165 Randomized Treatment LEV
Number analyzed (Participants) | 18 | 42
Percent change
  >= 1 d - <= 3 m: number analyzed (Participants) | 15 | 25
  >= 1 d - <= 3 m | -100.00 [-100.00 to -24.55] | -100.00 [-100.00 to -32.50]
  > 3 m - <= 6 m: number analyzed (Participants) | 12 | 24
  > 3 m - <= 6 m | -93.96 [-100.00 to -59.36] | -100.00 [-100.00 to -32.10]
  > 6 m - <= 9 m: number analyzed (Participants) | 11 | 22
  > 6 m - <= 9 m | -88.73 [-100.00 to 38.32] | -100.00 [-100.00 to -43.42]
  > 9 m - <= 12 m: number analyzed (Participants) | 11 | 22
  > 9 m - <= 12 m | -100.00 [-100.00 to -54.73] | -100.00 [-100.00 to -40.03]
  > 12 m - <= 15 m: number analyzed (Participants) | 11 | 18
  > 12 m - <= 15 m | -88.33 [-100.00 to -49.70] | -100.00 [-100.00 to -64.50]
  > 15 m - <= 18 m: number analyzed (Participants) | 11 | 18
  > 15 m - <= 18 m | -100.00 [-100.00 to -62.28] | -100.00 [-100.00 to -69.82]
  > 18 m - <= 21 m: number analyzed (Participants) | 9 | 17
  > 18 m - <= 21 m | -90.42 [-100.00 to -54.73] | -100.00 [-100.00 to -25.61]
  > 21 m - <= 24 m: number analyzed (Participants) | 9 | 16
  > 21 m - <= 24 m | -80.56 [-100.00 to -24.55] | -100.00 [-100.00 to -68.35]
  > 24 m - <= 27 m: number analyzed (Participants) | 9 | 15
  > 24 m - <= 27 m | -91.92 [-100.00 to -24.55] | -100.00 [-100.00 to -45.54]
  > 27 m - <= 30 m: number analyzed (Participants) | 9 | 15
  > 27 m - <= 30 m | -92.11 [-100.00 to -74.85] | -100.00 [-100.00 to -45.54]
  > 30 m - <= 33 m: number analyzed (Participants) | 8 | 15
  > 30 m - <= 33 m | -77.02 [-95.91 to 16.78] | -100.00 [-100.00 to -86.64]
  > 33 m - <= 36 m: number analyzed (Participants) | 8 | 13
  > 33 m - <= 36 m | -74.30 [-91.72 to -46.59] | -100.00 [-100.00 to -92.19]
  > 36 m - <= 39 m: number analyzed (Participants) | 8 | 13
  > 36 m - <= 39 m | -85.67 [-96.25 to -7.06] | -100.00 [-100.00 to -83.77]
  > 39 m - <= 42 m: number analyzed (Participants) | 7 | 10
  > 39 m - <= 42 m | -83.23 [-100.00 to -21.27] | -100.00 [-100.00 to -47.52]
  > 42 m - <= 45 m: number analyzed (Participants) | 6 | 7
  > 42 m - <= 45 m | -79.75 [-100.00 to -56.26] | -100.00 [-100.00 to -49.70]
  > 45 m - <= 48 m: number analyzed (Participants) | 4 | 7
  > 45 m - <= 48 m | -95.81 [-100.00 to -83.23] | -100.00 [-100.00 to -85.94]
  > 48 m - <= 51 m: number analyzed (Participants) | 4 | 6
  > 48 m - <= 51 m | -95.98 [-100.00 to -87.62] | -100.00 [-100.00 to -100.00]
  > 51 m - <= 54 m: number analyzed (Participants) | 4 | 4
  > 51 m - <= 54 m | -100.00 [-100.00 to -91.67] | -100.00 [-100.00 to -100.00]
  > 54 m: number analyzed (Participants) | 2 | 1
  > 54 m | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -100.00]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 1 (Week 0) until 2 weeks after termination (up to 54 months).
Description: Adverse events refer to the Full Analysis Set (FAS).
Groups:
- N165 Randomized Treatment PBO (FAS): Subjects received Placebo (PBO) in study N165 [NCT00600509] and received LEV in this study: After starting with the 4 week-fixed 3000 mg/day, the daily doses of LEV were permitted to be adjusted by 500 or 1000 mg/day at a 4-week interval between 1000 mg/day and 3000 mg/day. In the Placebo group the Serious Adverse Events (SAEs) Status epilepticus and Agitation occurred twice in 2 subjects.
Arm/Group | N165 Randomized Treatment PBO (FAS) | N165 Randomized Treatment LEV (FAS)
All-Cause Mortality (participants affected / at risk) | 0/50 | 1/101
Serious Adverse Events (participants affected / at risk) | 12/50 | 22/101
Other Adverse Events (participants affected / at risk) | 48/50 | 99/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N165 Randomized Treatment PBO (FAS) (N=50) | N165 Randomized Treatment LEV (FAS) (N=101)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Difficulty in walking (General disorders) | 1 | 0
Drowning (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Pyelonephritis acute (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Polytraumatism (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 5
Dyslalia (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 2 | 4
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0
Mass excision (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | N165 Randomized Treatment PBO (FAS) (N=50) | N165 Randomized Treatment LEV (FAS) (N=101)
Conjunctivitis (Eye disorders) | 3 | 2
Diplopia (Eye disorders) | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Abdominal pain upper (Gastrointestinal disorders) | 2 | 9
Cheilitis (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 4 | 20
Diarrhoea (Gastrointestinal disorders) | 5 | 27
Gastritis (Gastrointestinal disorders) | 4 | 6
Gingivitis (Gastrointestinal disorders) | 1 | 7
Nausea (Gastrointestinal disorders) | 6 | 13
Stomatitis (Gastrointestinal disorders) | 4 | 11
Toothache (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 5 | 13
Chest pain (General disorders) | 4 | 2
Malaise (General disorders) | 2 | 6
Pyrexia (General disorders) | 9 | 14
Seasonal allergy (Immune system disorders) | 3 | 4
Dental caries (Infections and infestations) | 6 | 13
Influenza (Infections and infestations) | 2 | 8
Nasopharyngitis (Infections and infestations) | 38 | 76
Pharyngitis (Infections and infestations) | 3 | 8
Arthropod sting (Injury, poisoning and procedural complications) | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 16 | 29
Excoriation (Injury, poisoning and procedural complications) | 9 | 18
Joint sprain (Injury, poisoning and procedural complications) | 5 | 8
Mouth injury (Injury, poisoning and procedural complications) | 2 | 6
Open wound (Injury, poisoning and procedural complications) | 4 | 6
Skin laceration (Injury, poisoning and procedural complications) | 5 | 14
Thermal burn (Injury, poisoning and procedural complications) | 2 | 10
Blood alkaline phosphatase increased (Investigations) | 3 | 3
Blood triglycerides increased (Investigations) | 3 | 6
Blood urine present (Investigations) | 3 | 2
Gamma-glutamyltransferase increased (Investigations) | 8 | 16
Glucose urine present (Investigations) | 3 | 6
Neutrophil count decreased (Investigations) | 0 | 8
Protein urine present (Investigations) | 5 | 3
Weight decreased (Investigations) | 3 | 9
Weight increased (Investigations) | 2 | 7
White blood cell count increased (Investigations) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 8
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Convulsion (Nervous system disorders) | 2/5 | 9
Dizziness (Nervous system disorders) | 12 | 20
Epilepsy (Nervous system disorders) | 2 | 6
Headache (Nervous system disorders) | 16 | 28
Hypoaesthesia (Nervous system disorders) | 4 | 4
Migraine (Nervous system disorders) | 4 | 1
Somnolence (Nervous system disorders) | 13 | 25
Tremor (Nervous system disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 8 | 13
Pollakiuria (Renal and urinary disorders) | 3 | 5
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 12 | 22
Acne (Skin and subcutaneous tissue disorders) | 2 | 8
Eczema (Skin and subcutaneous tissue disorders) | 5 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days